CLINICAL TRIAL: NCT05878977
Title: Effectiveness of Immunotherapy in the First-line Treatment of Disseminated Melanoma and Recognition of Prognostic and Predictive Biomarkers From the Primary Tumor, Stool and Body Fluids: PROTOCOL TRIAL
Brief Title: Biomarkers in Immunotherapy of Melanoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Oncology Ljubljana (Other)
Collaborators: Blood Transfusion Centre of Slovenia (Other Government); University Medical Centre Ljubljana (Other); University of Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERIDNPVO-0034/2021
Record Dates: First submitted 2023-04-19; First posted 2023-05-30 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Melanoma; Immune Checkpoints Inhibitors; Gastrointestinal Microbiome (Bacterial and Viral); Exosomal mRNA Expression of PD-L1 and IFNγ
MeSH Terms: conditions — Melanoma | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Immune checkpoint inhibitors (Other)
  Interventions: Drug: Immune checkpoint inhibitor

INTERVENTIONS:
Drug: Immune checkpoint inhibitor — Identification of novel predictive and prognostic biomarkers for immunotherapy treatment response in metastatic melanoma

SUMMARY:
Background: Immunotherapy has been successful in treating advanced melanoma, but a large proportion of patients do not respond to the treatment with immune checkpoint inhibitors (ICIs). Preclinical and small cohort studies suggest biomarkers from the primary tumor, stool and body fluids as markers of response. This prospective study will evaluate gastrointestinal microbiome (bacterial spices and virome) composition and exosomal mRNA expression of PD-L1 and IFNγ correlation with radiological response rates to ICIs treatment of advanced melanoma patients. Methods: Patients treated with immune checkpoint inhibitors as a first line treatment for metastatic melanoma are recruted to the study. Stool samples are submitted before the start of treatment, at the 12 (+/-2) week and 28 (+/-4) week, and at the event ( such as, suspected disease progression/hyperprogressio, immune related adverse event (irAE), etc). Peripheral venous blood samples are taken additionaly at the same time points for cytologic and molecular tests. Histological material from the tumor tissue is obtained before the start of immunotherapy treatment. Primary objectives are to determine whether human gastrointestinal microbiome (bacterial and viral) and exosomal mRNA expression of PD-L1 and IFNγ predict response to treatment with PD-1 and CTLA-4 inhibitors and are associated with occurrence of irAE in patients with metastatic melanoma at different time points. Response is evaluated radiologically with imaging methods in accordance with the irRECIST criteria. Conclussion: Despite the great success of the treatment of metastatic melanoma with immunotherapy, there remains a significant proportion of patients who do not respond to treatment or who develop severe adverse events during treatment. Identification of novel predictive and prognostic biomarkers for immunotherapy treatment response is therefore necessary. This study is the first to combine and investigate multiple potential predictive and prognostic biomarkers and its dynamics. The results could serve for a better and multi-level understanding of the various factors influencing immunotherapy treatment.

DETAILED DESCRIPTION:
The goal of this [type of study: observational study or clinical trial] is to [learn about, test, compare etc.] in [describe participant population/health conditions]. The main question[s] it aims to answer are:

* [question 1]
* [question 2] Participants will [describe the main tasks participants will be asked to do, treatments they'll be given and use bullets if it is more than 2 items].

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Cytologically or histologically verified malignant melanoma
* Stage IIID unresectable/IV according to AJCC classification (8th edition, 2018)
* Performance status according to WHO 0 - 2 (ECOG criteria)
* 1st line of systemic treatment with immunotherapy (nivolumab, ipi/nivo, pembrolizumab)
* Triple CT/PET CT done within 4 weeks before the first application
* Signed consent to participate in clinical research

Exclusion Criteria:

* Previously treated melanoma with systemic therapy
* Capacity status according to WHO 3 - 4 (ECOG criteria)
* Contraindications for immunotherapy treatment (known deficiency of the immune system or active immunosuppressive treatment or active autoimmune disease requiring treatment)
* Other malignant diseases (except cured basal cell carcinoma and squamous cell carcinoma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
response prediction in first line immune checkpoint inhibitors treatment in metastatic melanoma assessed by human gastrointestinal microbiome (bacterial and viral) and exosomal mRNA expression of PD-L1 and IFNγ | 3 years
  Primary objectives are to determine whether human gastrointestinal microbiome (bacterial and viral) and exosomal mRNA expression of PD-L1 and IFNγ predicts response to treatment with PD-1 and CTLA-4 inhibitors and are associated with occurrence of irAE in patients with metastatic melanoma.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Oncology Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided